CLINICAL TRIAL: NCT02550093
Title: The Effect of Intranasal Oxytocin on Pain Sensitivity and Threshold: A Randomized, Double Blinded, Crossover Volunteer Study
Brief Title: The Effect of Intranasal Oxytocin on Pain Sensitivity and Threshold
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Walega, Associate Professor, Chief, Division of Pain Medicine, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: STU86297
Record Dates: First submitted 2015-04-16; First posted 2015-09-15 (Estimated); Results first posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Healthy
Keywords: Volunteers
MeSH Terms: interventions — tioconazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin, then Normal Saline (Experimental): Each subject will receive nasal spray(s) into each nostril of 4 Units up to 32 units of Oxytocin prior to Thermal Evaluation System Testing on intervention 1 (day 1). Following a wash-out period of 13 days the same subject will then receive a nasal spray(s) into each nostril of 4 Units up to 32 units of Normal Saline prior to Thermal Evaluation System Testing on intervention 2 (day 14).
  Interventions: Procedure: Intervention 1; Behavioral: Washout Period; Procedure: Intervention 2
- Normal Saline, then Oxytocin (Experimental): Each subject will receive nasal spray(s) into each nostril of 4 Units up to 32 units of Normal Saline prior to Thermal Evaluation System Testing on intervention 1 (day 1). Following a wash-out period of 14 to 15 days the same subject will then receive nasal spray(s) into each nostril of 4 Units up to 32 units of Oxytocin prior to Thermal Evaluation System Testing on intervention 2 (day 14).
  Interventions: Procedure: Intervention 1; Behavioral: Washout Period; Procedure: Intervention 2

INTERVENTIONS:
Procedure: Intervention 1 — Each subject will receive nasal spray(s) into each nostril of 4 Units up to 32 units of study drug prior to Thermal Evaluation System Testing on intervention 1 (Day 1).
  Other Names: Day 1
Behavioral: Washout Period — The wash-out period will be between intervention 1 and intervention 2. 13 days in length.
Procedure: Intervention 2 — Each subject will receive nasal spray(s) into each nostril of 4 Units up to 32 units of study drug prior to Thermal Evaluation System Testing on intervention 2 (Day 14).
  Other Names: Day 14

SUMMARY:
Oxytocin is neurohypophysial peptide that acts mainly as a neuromodulator in the brain.The vast majority of basic science studies suggested a large effect of oxytocin in minimizing acute pain.Few studies have demonstrated an association between plasma levels of oxytocin and pain in humans. Since addictive properties of oxytocin have not been described, the drug may have important application in the management of acute and chronic pain. No studies have examined the effect of intranasal oxytocin on pain sensitivity and threshold.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females volunteers, English speaking

Exclusion Criteria:

* Pregnancy, lactation, allergy to preservatives, mental disease, any chronic pain and any current use of analgesics, anxiety or depression.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Walega, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yamasue H, Yee JR, Hurlemann R, Rilling JK, Chen FS, Meyer-Lindenberg A, Tost H. Integrative approaches utilizing oxytocin to enhance prosocial behavior: from animal and human social behavior to autistic social dysfunction. J Neurosci. 2012 Oct 10;32(41):14109-17. doi: 10.1523/JNEUROSCI.3327-12.2012. PMID 23055480
- [Background] Fewtrell MS, Loh KL, Blake A, Ridout DA, Hawdon J. Randomised, double blind trial of oxytocin nasal spray in mothers expressing breast milk for preterm infants. Arch Dis Child Fetal Neonatal Ed. 2006 May;91(3):F169-74. doi: 10.1136/adc.2005.081265. Epub 2005 Oct 13. PMID 16223754
- [Background] MacDonald E, Dadds MR, Brennan JL, Williams K, Levy F, Cauchi AJ. A review of safety, side-effects and subjective reactions to intranasal oxytocin in human research. Psychoneuroendocrinology. 2011 Sep;36(8):1114-26. doi: 10.1016/j.psyneuen.2011.02.015. Epub 2011 Mar 23. PMID 21429671
- [Background] Rash JA, Aguirre-Camacho A, Campbell TS. Oxytocin and pain: a systematic review and synthesis of findings. Clin J Pain. 2014 May;30(5):453-62. doi: 10.1097/AJP.0b013e31829f57df. PMID 23887343
- [Background] Wang YL, Yuan Y, Yang J, Wang CH, Pan YJ, Lu L, Wu YQ, Wang DX, Lv LX, Li RR, Xue L, Wang XH, Bi JW, Liu XF, Qian YN, Deng ZK, Zhang ZJ, Zhai XH, Zhou XJ, Wang GL, Zhai JX, Liu WY. The interaction between the oxytocin and pain modulation in headache patients. Neuropeptides. 2013 Apr;47(2):93-7. doi: 10.1016/j.npep.2012.12.003. Epub 2013 Jan 30. PMID 23375440
- [Background] Singer T, Snozzi R, Bird G, Petrovic P, Silani G, Heinrichs M, Dolan RJ. Effects of oxytocin and prosocial behavior on brain responses to direct and vicariously experienced pain. Emotion. 2008 Dec;8(6):781-91. doi: 10.1037/a0014195. PMID 19102589

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cross-over study design
Period: Intervention 1
Arm/Group | Oxytocin, Then Normal Saline | Normal Saline, Then Oxytocin
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Wash-out Period
Arm/Group | Oxytocin, Then Normal Saline | Normal Saline, Then Oxytocin
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Intervention 2
Arm/Group | Oxytocin, Then Normal Saline | Normal Saline, Then Oxytocin
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Volunteers
Groups:
- All Study Participants: Each subject will receive nasal spray(s) into each nostril of 4 Units up to 32 units of either Oxytocin then Normal Saline or Normal Saline then Oxytocin prior to Thermal Evaluation System Testing.
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 24 [22 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Hot and Cold Thermal Sensory Threshold for Pain at Baseline in Degrees Celsius.
Description: Thermal Sensory Threshold for Pain at baseline prior to study drug administration. Evaluation of subjects baseline responses of perception of hot and cold stimuli utilizing the Medoc Pathway Pain &Sensory Evaluation System (Medoc Ltd, Israel). The baseline response variable was estimated by averaging the subjects response over three trials, with an interval of 30 seconds. A thermode was attached to the subjects hand and the subject was asked to press a mouse button when they perceive the sensation of heat pain or cold pain. The temperature range was 51C to 0C.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: degrees Celsius
Groups:
- Oxytocin; Normal Saline: Baseline recording - no study drug administerd prior to Thermal Evaluation System Testing.
Arm/Group | Oxytocin | Normal Saline
Number analyzed (Participants) | 20 | 20
degrees Celsius
  Heat | 43.93 (4.18) | 43.0 (4.34)
  Cold | 14.81 (11.10) | 13.33 (10.51)
Statistical Analysis 1: Comparison: Oxytocin vs Normal Saline; HEAT; Test type: Superiority or Other; p = .47, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Oxytocin vs Normal Saline; COLD; Test type: Superiority or Other; p = 0.70, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Hot and Cold Thermal Sensory Threshold for Pain at 45 Minutes in Degrees Celsius.
Description: Thermal Sensory Threshold for Pain at 45 minutes after study drug administration. Evaluation of subjects responses of perception of hot and cold stimuli utilizing the Medoc Pathway Pain &Sensory Evaluation System (Medoc Ltd, Israel). The response variable was estimated by averaging the subjects response over three trials, with an interval of 30 seconds. A thermode was attached to the subjects hand and the subject was asked to press a mouse button when they perceive the sensation of heat pain or cold pain. The temperature range was 51C to 0C.
Time Frame: 45 minutes
Measure: Mean (Standard Deviation); unit: degrees Celsius
Groups:
- Oxytocin: Each subject will receive nasal spray(s) into each nostril of 4 Units up to 32 units of Oxytocin prior to Thermal Evaluation System Testing.
  Oxytocin: Each subject will receive nasal spray(s) into each nostril of 4 Units up to 32 units of study drug prior to Thermal Evaluation System Testing.
- Normal Saline: Each subject will receive nasal spray(s) into each nostril of 4 Units up to 32 units of Normal Saline prior to Thermal Evaluation System Testing.
  Normal Saline: Each subject will receive nasal spray(s) into each nostril of 4 Units up to 32 units of study drug prior to Thermal Evaluation System Testing.
Arm/Group | Oxytocin | Normal Saline
Number analyzed (Participants) | 20 | 20
degrees Celsius
  Heat | 43.60 (3.68) | 43.42 (3.98)
  Cold | 15.68 (10.60) | 15.17 (10.88)
Statistical Analysis 1: Comparison: Oxytocin vs Normal Saline; HEAT; Test type: Superiority or Other; p = 0.84, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Oxytocin vs Normal Saline; COLD; Test type: Superiority or Other; p = 0.95, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Hot and Cold Thermal Sensory Threshold for Pain at 90 Minutes in Degrees Celsius.
Description: Thermal Sensory Threshold for Pain at 90 minutes after study drug administration. Evaluation of subjects responses of perception of hot and cold stimuli utilizing the Medoc Pathway Pain &Sensory Evaluation System (Medoc Ltd, Israel). The response variable was estimated by averaging the subjects response over three trials, with an interval of 30 seconds. A thermode was attached to the subjects hand and the subject was asked to press a mouse button when they perceive the sensation of heat pain or cold pain. The temperature range was 51C to 0C.
Time Frame: 90 minutes
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Oxytocin | Normal Saline
Number analyzed (Participants) | 20 | 20
degrees Celsius
  Heat | 43.94 (3.97) | 43.95 (3.80)
  Cold | 15.41 (11.24) | 12.96 (11.38)
Statistical Analysis 1: Comparison: Oxytocin vs Normal Saline; HEAT; Test type: Superiority or Other; p = 0.92, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Oxytocin vs Normal Saline; COLD; Test type: Superiority or Other; p = 0.63, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Mechanical Pain Threshold for Pain at Baseline in Grams.
Description: Mechanical pain threshold for pain at baseline utilizing a digital electrovonfrey anesthesiometer (IITC model Alemo 2290-4; Woodland Hills, CA, USA). The subjects response to painful stimulus was recorded in grams. Each variable was estimated by averaging a participant's responses over 3 trials, with an intertrial interval of 30 s. The lower amount in grams the more sensitive you are to pain.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Oxytocin | Normal Saline
Number analyzed (Participants) | 20 | 20
Grams | 194.90 (117.52) | 223.31 (149.56)
Statistical Analysis 1: Comparison: Oxytocin vs Normal Saline; Test type: Superiority or Other; p = 0.60, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Mechanical Pain Threshold for Pain at 45 Minutes in Grams.
Description: Mechanical pain threshold for pain at 45 minutes utilizing a digital electrovonfrey anesthesiometer (IITC model Alemo 2290-4; Woodland Hills, CA, USA). The subjects response to painful stimulus was recorded in grams. Each variable was estimated by averaging a participant's responses over 3 trials, with an intertrial interval of 30 s. The lower amount in grams the more sensitive you are to pain.
Time Frame: 45 minutes
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Oxytocin | Normal Saline
Number analyzed (Participants) | 20 | 20
Grams | 195.07 (145.41) | 197.49 (124.71)
Statistical Analysis 1: Comparison: Oxytocin vs Normal Saline; Test type: Superiority or Other; p = 0.68, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Mechanical Pain Threshold for Pain at 90 Minutes in Grams.
Description: Mechanical pain threshold for pain at 90 minutes utilizing a digital electrovonfrey anesthesiometer (IITC model Alemo 2290-4; Woodland Hills, CA, USA). The subjects response to painful stimulus was recorded in grams. Each variable was estimated by averaging a participant's responses over 3 trials, with an intertrial interval of 30 s. The lower amount in grams the more sensitive you are to pain.
Time Frame: 90 minutes
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Oxytocin | Normal Saline
Number analyzed (Participants) | 20 | 20
Grams | 198.76 (141.41) | 208.77 (124.97)
Statistical Analysis 1: Comparison: Oxytocin vs Normal Saline; Test type: Superiority or Other; p = 0.62, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Suprathreshold Magnitude for Pain at Baseline Measured in Visual Analog Pain Scores.
Description: Supra-threshold magnitude for pain was assessed utilizing the Medoc Pathway System with contact heat evoked potential simulator at 49 degrees Celsius. Visual analog pain score ranges from 0 (no pain) to 10 (worst pain imaginable).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Oxytocin | Normal Saline
Number analyzed (Participants) | 20 | 20
scores on a scale | 2.90 (1.65) | 3.02 (1.88)
Statistical Analysis 1: Comparison: Oxytocin vs Normal Saline; Test type: Superiority or Other; p = 0.97, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Suprathreshold Magnitude for Pain at 45 Minutes Measured in Visual Analog Pain Scores.
Description: as for outcome 7
Time Frame: 45 minutes
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Oxytocin | Normal Saline
Number analyzed (Participants) | 20 | 20
scores on a scale | 2.58 (1.37) | 2.67 (1.59)
Statistical Analysis 1: Comparison: Oxytocin vs Normal Saline; Test type: Superiority or Other; p = 0.97, Wilcoxon (Mann-Whitney)

9. Primary Outcome: Suprathreshold Magnitude for Pain at 90 Minutes Measured in Visual Analog Pain Scores.
Description: as for outcome 7
Time Frame: 90 minutes
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Oxytocin | Normal Saline
Number analyzed (Participants) | 20 | 20
scores on a scale | 2.53 (1.58) | 2.29 (1.51)
Statistical Analysis 1: Comparison: Oxytocin vs Normal Saline; Test type: Superiority or Other; p = 0.61, Wilcoxon (Mann-Whitney)

10. Primary Outcome: Thermal Wind-up Pain Assessment at Baseline
Description: Using a Visual Analog Scale (VAS) subjects will be asked to rate the painfulness of the stimulus for thermal wind-up pain utilizing the medoc pathway system. Each VAS score was recorded over 10 trials, with an interval of 3s. The average VAS score was reported. Visual analog scale ranges from 0 (no pain) to 10 (worst pain imaginable).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Oxytocin | Normal Saline
Number analyzed (Participants) | 20 | 20
scores on a scale | 3.59 (2.09) | 3.15 (1.90)
Statistical Analysis 1: Comparison: Oxytocin vs Normal Saline; Test type: Superiority or Other; p = 0.71, Wilcoxon (Mann-Whitney)

11. Primary Outcome: Thermal Wind-up Pain at 45 Minutes
Description: as for outcome 10
Time Frame: 45 minutes
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Oxytocin | Normal Saline
Number analyzed (Participants) | 20 | 20
scores on a scale | 2.99 (1.71) | 2.85 (1.92)
Statistical Analysis 1: Comparison: Oxytocin vs Normal Saline; Test type: Superiority or Other; p = 0.74, Wilcoxon (Mann-Whitney)

12. Primary Outcome: Thermal Wind-up Pain at 90 Minutes
Description: as for outcome 10
Time Frame: 90 minutes
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Oxytocin | Normal Saline
Number analyzed (Participants) | 20 | 20
scores on a scale | 2.82 (1.63) | 2.63 (1.66)
Statistical Analysis 1: Comparison: Oxytocin vs Normal Saline; Test type: Superiority or Other; p = 0.75, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 24hrs after intervention.
Description: Assessments completed 24 hours after participants who completed study interventions.
Groups:
- Oxytocin: Subjects received nasal spray(s) into each nostril of 4 Units up to 32 units of Oxytocin prior to Thermal Evaluation System Testing.
- Normal Saline: Subjects received nasal spray(s) into each nostril of Normal Saline prior to Thermal Evaluation System Testing.
Arm/Group | Oxytocin | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
Though we used the same method of intranasal administration as preceding studies, it is possible that the oxytocin did not reach peak levels at the time of the testing or was not absorbed. We did not assess plasma levels of oxytocin to assess whether absorption occurred and was consistent among all participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes